CLINICAL TRIAL: NCT03525353
Title: Comparison Of Radiation Exposure To Patients During ERCPs Performed By Endoscopists Trained In Judicious Use Of Fluoroscopy With Those Without Formal Training
Brief Title: Comparison Of Radiation Exposure To Patients During Endoscopic Retrograde Cholangiopancreatography (ERCP) Performed By Endoscopists Trained In Judicious Use Of Fluoroscopy With Those Without Formal Training
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Nirav C Thosani, Assistant Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-15-0019
Record Dates: First submitted 2016-01-04; First posted 2018-05-15 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients undergoing ERCP by formally trained Endoscopists: Patients who undergo ERCP (Endoscopic Retrograde Cholangio Pancreatography) performed by Endoscopists who are trained on minimum use of fluoroscopy.
  Interventions: Other: Endoscopic retrograde cholangiopancreatography - No Intervention have been used other than standard of care
- Patients undergoing ERCP by Endoscopists not formally trained: Patients who undergo ERCP (Endoscopic Retrograde Cholangio Pancreatography) performed by Endoscopists who have not received formal training on minimum use of fluoroscopy.
  Interventions: Other: Endoscopic retrograde cholangiopancreatography - No Intervention have been used other than standard of care

INTERVENTIONS:
Other: Endoscopic retrograde cholangiopancreatography - No Intervention have been used other than standard of care — No intervention has been used and this is an observational study

SUMMARY:
Purpose: To compare the radiation exposure in patients during Endoscopic retrograde cholangiopancreatography (ERCP) done by Endoscopists formally trained in judicious use of fluoroscopy versus ERCPs done by Endoscopists without such formal training.

Research design: This is an observational study to compare radiation exposure in patients during ERCPs based on formal training.

Procedures to be used: None Risks and potential benefits There are no risks associated with this study as it is a retrospective chart review. Potential benefits include the knowledge gained from this study which may be of help to patients in the future.

Importance of knowledge that may reasonably be expected to result The knowledge gained from this study may be of help to provide new insights and develop newer guidelines for radiation use in the future.

ELIGIBILITY:
Inclusion Criteria:

* Any indications for undergoing an ERCP. If a patient undergoes more than one ERCP then it shall be reported as such, as multiple data points.
* Only those ERCP cases will be included that have been exposed to fluoroscopy (X-ray radiation).
* Adult populations will be included, all races and belonging to any gender will be included in the study.

Exclusion Criteria:

* Patients who didn't receive ERCP
* Those in whom the biliary or pancreatic ducts are not cannulated and therefore who do not receive any fluoroscopy
* Pregnant women
* Patient population less than 18 years of age

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Any indications for undergoing an ERCP. If a patient undergoes more than one ERCP then it shall be reported as such, as multiple data points.
  Only those ERCP cases will be included that have been exposed to fluoroscopy (X-ray radiation).
  Those in whom the biliary or pancreatic ducts are not cannulated and therefore who do not receive any fluoroscopy will be excluded.
  Adult populations will be included, all races and belonging to any gender will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-11; Primary Completion 2021-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Radiation exposure as assessed by fluoroscopy time | at the time of ERCP
  Radiation exposure of patients who undergo ERCP (Endoscopic Retrograde Cholangio Pancreatography) will be assessed by fluoroscopy time, which is indicated by the device used for ERCP. Fluoroscopy time at the time of ERCP will be recorded at the end of the procedure and is documented by the endoscopy technician.
Radiation exposure as assessed by total emittance | at the time of ERCP
  Radiation exposure of patients who undergo ERCP (Endoscopic Retrograde Cholangio Pancreatography) will be assessed by total emittance, which is indicated by the device used for ERCP. Total emittance at the time of ERCP will be recorded at the end of the procedure and is documented by the endoscopy technician.

CONTACTS AND LOCATIONS:
Overall Officials: Nirav Thosani, MD MHA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States